CLINICAL TRIAL: NCT06793553
Title: Randomized Phase II Trial Evaluating the Efficacy of Paclitaxel+Bevacizumab INDUCtion Followed by at atEzolizumab+Nab-paclitaxel for PD-L1-positive Metastatic Triple Negative Breast Cancer (JBCRG-M10, CMA-0196) (INDUCE Trial)
Brief Title: Induction Therapy of PTX+BV Followed by Atezolizumab+Nab-PTX for PD-L1+ TNBC
Acronym: INDUCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Breast Cancer Research Group (Other)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBCRG-M10
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
Keywords: PD-L1-positive; bevacizumab; induction therapy; immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction therapy group (Active Comparator): 2 cycles of PTX + bevacizumab → atezolizumab + nab-PTX
  Interventions: Drug: Induction therapy
- Control group (standard treatment group) (Experimental): Atezolizumab + nab-PTX
  Interventions: Drug: Induction therapy

INTERVENTIONS:
Drug: Induction therapy — 2 cycles of PTX+ bevacizumab induction therapy followed by atezolizumab+nab-PTX

SUMMARY:
The objective of this research is to evaluate the efficacy of the treatment strategy to administer atezolizumab + nab-paclitaxel (PTX) following 2 cycles of induction therapy with PTX + bevacizumab (induction treatment strategy) in programmed cell death ligand-1 (PD-L1)-positive metastatic triple-negative breast cancer (mTNBC) in comparison with the standard atezolizumab + nab-PTX therapy.

DETAILED DESCRIPTION:
The objective of this research is to evaluate the efficacy of the treatment strategy to administer atezolizumab + nab-PTX following 2 cycles of induction therapy with PTX + bevacizumab (induction treatment strategy) in PD-L1-positive mTNBC in comparison with the standard atezolizumab + nab-PTX therapy in a rondomized phase II design.

It is hypothesized in this research that in patients with PD-L1-positive mTNBC, 2 cycles of PTX+ bevacizumab induction therapy induce early response and an immune microenvironment conducive to the benefits of immunotherapy, and improve progression-free survival as compared with the standard treatment with atezolizumab + nab-PTX therapy (standard treatment group). The primary objective of this research is to investigate this hypothesis.

A key secondary objective is to compare the 2-year PFS rate between the induction therapy group and the standard treatment group in order to assess the long-term effect of the induction treatment strategy. Furthermore, in patients in the induction therapy group who are not assessed as PD in the first imaging assessment, the 2-year PFS rate will be compared to the reference value expected in a historical control to examine the benefits of the induction therapy.

Other secondary objectives are to compare the response rate and the disease control rate as efficacy endpoints and to evaluate the effect of the induction treatment strategy on early PD. Overall survival (OS) will also be compared.

In addition, with the aim of exploring the mechanism by which the induction treatment strategy contributes to enhancement of the effect of the standard treatment with atezolizumab + nab-PTX therapy, the immune status in the tumor microenvironment and peripheral blood will be evaluated, and its relationship with antitumor effects will be investigated.

For evaluation of efficacy and safety in the induction therapy group, 2 cycles of induction therapy + immunochemotherapy will be evaluated as a series of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with metastatic recurrent or unresectable advanced TNBC
2. Documented PD-L1 positivity (SP142 IC ≥ 1) confirmed by local assessment of the most recent tumor sample or an archival tumor sample.
3. In the case of patients who were candidates for curative treatment, the duration from the completion of the curative treatment {date of surgery for primary breast cancer or date of last dose of peri-operative drug therapy (including anthracycline regimen, taxane regimen, anti-PD-(L)1 antibody, capecitabine, poly ADP-ribose polimerase [PARP] inhibitors, etc.), whichever is later} to the first local or distant recurrence should be at least 6 months. The date of postoperative radiotherapy is not included in this calculation. The use of anti-PD-(L)1 antibodies is allowed during perioperative drug therapy.
4. ECOG PS 0-1
5. Female or male aged 18 years or older.
6. Histologically or cytologically confirmed TNBC that is ER-negative (< 10% positive cell occupancy or Allred Proportion score of 0-2), HER2-negative (IHC 1+ or less or FISH/DISH negative) according to ASCO/CAP Criteria 2018 (in the case of IHC2+, negativity is confirmed by FISH/DISH).
7. Patients who have not received chemotherapy for metastatic recurrent or unresectable advanced cancer. However, prior treatment with PARP inhibitors for metastatic recurrent or unresectable advanced cancers in patients with pathogenic BRCA variants is allowed.
8. Having measurable or non-measurable lesions as assessed by local CT or MRI. Tumor lesions located at a previously irradiated site will be considered evaluable if unequivocal progression is seen after radiation.
9. Laboratory tests performed within 14 days before enrollment meet the following criteria [1] to [8]. However, patients must not have received granulocyte colony-stimulating factor (G-CSF) or blood transfusion within 14 days prior to the date of blood sampling.

[1] Neutrophil count ≥ 1500/mm3 [2] Platelet count ≥ 10 x 104/mm3 [3] Hemoglobin ≥ 8.0 g/dL [4] AST (GOT) ≤ 100 IU/L (≤ 200 IU/L if liver metastasis is present) [5] ALT (GPT) ≤ 100 IU/L(≤ 200 IU/L if liver metastasis is present) [6] Total bilirubin ≤ 1.5 mg/dL Total bilirubin < 3.0 mg/dL for patients with Gilbert's syndrome [7] Creatinine ≤ 1.5 mg/dL [8] Any of the following criteria is met: i) Urine protein (dipstick) is negative (-) or 1+ ii) If urine protein (dipstick) is ≥ 2+; Measurement of 24-hour urine protein shows urine protein ≤ 1 g/24 hours (may be substituted by urine protein/creatinine ratio ≤ 1)

(10) Blood pressure is sufficiently controlled (systolic blood pressure ≤ 150 mmHg and diastolic blood pressure ≤ 90 mmHg with ≤ 2 antihypertensive drugs [counted as the number of combinations]).

(11) Patients expected to survive for at least 3 months.

(12) Written consent has been obtained from the patient himself/herself after sufficient explanation of the contents of the study before registration.

(13) In the case of female patients of childbearing potential (including patients who have no menstruation for medical reasons such as chemical menopause), the patients must agree to continue to practice contraception until 5 months after the last dose of atezolizumab or 6 months after the last dose of bevacizumab, nab-PTX or PTX, whichever comes later. Patients must also agree not to breastfeed during study treatment and for at least 5 months after the last dose of atezolizumab and at least 6 months after the last dose of bevacizumab. In the case of male patients with a partner of childbearing potential, the patient whose partner must agree to continue to practice contraception until 6 months after the last administration of PTX and nab-PTX.

Exclusion Criteria:

1. Having active brain metastases or carcinomatous meningitis. Previously treated brain metastases are allowed if neurological symptoms have returned to baseline and are clinically stable for at least 2 weeks prior to enrollment.
2. Patients with a history of invasive malignancy within 3 years prior to enrollment. However, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or lesions equivalent to carcinoma in situ or intramucosal carcinoma that are assessed as cured by local treatment are not included in active double cancer.
3. Concurrent or metachronous bilateral invasive breast cancer. However, the patients will be accepted if bilateral lesions are TNBC and are confirmed to be PD-L1-positive by evaluation using a sample of a recurrent lesion.
4. Patients who have received radiotherapy within 14 days prior to enrollment. (Administration or irradiation on the same day of the week 14 days prior to the day of enrollment is permitted.)
5. Patients who have received other study drugs within 14 days prior to enrollment. (Administration on the same day of the week 14 days prior to the day of enrollment is permitted.)
6. Administration of a live vaccine within 30 days of the first dose of the study drug. Administration of inactivated vaccines is permitted.
7. Patients who have received systemic corticosteroid or immunosuppressant equivalent to prednisone exceeding 10 mg/day within 14 days prior to enrollment for active autoimmune disease. (excluding temporary administration for examination or prophylactic administration)
8. Active infection requiring systemic treatment.
9. Patients who concurrently have interstitial lung disease/pneumonitis at the time of enrollment or who have a history of interstitial lung disease/pneumonitis requiring systemic corticosteroids administration. (A history of radiation pneumonitis [fibrosis] within the radiation field is permitted.)
10. Patients who are pregnant, possibly pregnant, or lactating.
11. Patients who are positive for HBs antigen or HCV antibody. Patients positive for HCV antibody whose HCV virus level is below the detection limit will be permitted.
12. Patients who are positive for HIV-1 antibody or HIV-2 antibody (test is not essential for enrollment).
13. Patients with significant cardiovascular disease. Patients with a history of myocardial infarction, acute coronary artery disease, coronary angioplasty/stenting/bypass grafting within the last 6 months. Patients with congestive heart failure of Class III to IV of the New York Heart Association.
14. Patients with the following history/concomitant diseases:

[1] Poorly controlled diabetes mellitus [2] Grade ≥ 2 peripheral sensory neuropathy [3] Congenital haemorrhagic diathesis/coagulopathy [4] Arterial thromboembolism (cerebral infarction, etc.) or venous thromboembolism (deep vein thrombosis, pulmonary embolism, etc.) within 6 months prior to enrollment [5] Gastrointestinal perforation, active gastrointestinal ulcer, and Grade ≥ 3 haemorrhage (site not specified) [6] Other serious complications (renal failure, hepatic failure, etc.)

(15) Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's completion of the study, or is not in the best interest of the participant to participate in.

(16) Patients with any psychiatric condition that may interfere with the conduct of the study.

(17) Patients with a history of hypersensitivity to the study drug or its analogues.

(18) Patients with alcohol intolerance or a history of hypersensitivity to Cremophor.

(19) Patients with a history of active tuberculosis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) * | 2 years
  Whether the PFS is prolonged with statistical significance (level of significance, one-sided 10%) in the induction therapy group compared to the standard treatment group will be evaluated.
  * In this research, all antitumor effects will be assessed based on the evaluation by the primary physician.

SECONDARY OUTCOMES:
(1) 2-year PFS rate (2) 2-year PFS rate in patients with non-PD on the first imaging assessment in the induction therapy group | 2 years
  The standard treatment group and the induction therapy group will be compared and evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Yukinori Ozaki, Koto-ku, 3-8-31, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided